CLINICAL TRIAL: NCT05680441
Title: Evaluation of Annexin-A1, Carbonic Anhydrase-1, and Elongation Factor-1 Gamma Levels in Periodontal Diseases
Brief Title: GCF Annexin-A1, Carbonic Anhydrase-1, and Elongation Factor-1 Gamma Levels in Periodontitis
Status: Completed | Type: Observational
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Bilge Cansu UZUN SAYLAN, Assistant Prof, Dokuz Eylul University
Other Study IDs: CANSU35
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Periodontitis; Periodontal Inflammation
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Gingival crevicular fluid
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healty group: The controls/Healthy group were the individuals with well-maintained oral hygiene without no periodontal disease history or symptoms with a probing pocket depth (PPD) of ≤3 mm and bleeding on probing (BOP) of (+) ≤10.
  Interventions: Other: Peirodontal clinical measurements and gingival crevicular fluid sampling
- Periodontitis stage 3 grade B: Stage III periodontitis patients had at least 4 interdental sites clinical attachment level (CAL)> 5 mm due to periodontitis, radiographic bone loss reaching to the mid-third of the root or beyond, teeth loss less than 4 teeth due to periodontitis. These patients were graded according to the bone loss%/age index (Grade B, 0.25-1.00).
  Interventions: Other: Peirodontal clinical measurements and gingival crevicular fluid sampling
- Periodontitis stage 3 grade C: Stage III periodontitis patients had at least 4 interdental sites clinical attachment level (CAL)> 5 mm due to periodontitis, radiographic bone loss reaching to the mid-third of the root or beyond, teeth loss less than 4 teeth due to periodontitis.Since the bone loss (%)/age values were >1.0, all periodontitis patients were considered grade C.
  Interventions: Other: Peirodontal clinical measurements and gingival crevicular fluid sampling
- Gingivitis: Only generalized gingivitis patients were included in this study. Individuals presenting with a BOP≥30% and PPD≤3 mm without radiographic bone loss and attachment loss were considered to have gingivitis.
  Interventions: Other: Peirodontal clinical measurements and gingival crevicular fluid sampling

INTERVENTIONS:
Other: Peirodontal clinical measurements and gingival crevicular fluid sampling — The clinical periodontal examination of the healthy and periodontitis subjects consisted of plaque index (PI), probing pocket depth (PPD), clinical attachment level (CAL), and bleeding on probing (BOP) recorded. CAL was calculated by adding GR to the PPD values. Averages for full mouth PPD, CAL, and the percentage of sites with BOP were calculated for each subject. A single calibrated examiner (VO) conducted a full mouth periodontal examination of all participants.

SUMMARY:
The study aimed to investigate gingival crevicular fluid (GCF) levels of possible novel biomarkers Annexin-A1 (ANX A1), Carbonic anhydrase- 1 (CA I), and Elongation Factor-1 Gamma (EF1-Ɣ) in health along with different periodontal diseases.

In total, 80 systemically healthy individuals were included in this study; 20 with periodontitis stage 3 grade B , 20 with periodontitis stage 3 grade C (P-Stage III/C), 19 with gingivitis, and 21 with clinically healthy periodontium. Probing depth, clinical attachment level, plaque index, and papillary bleeding index were recorded. GCF ANX A1, CA I and EF1-Ɣ levels were analyzed by enzyme-linked immunosorbent assay (ELISA). Receiver operating characteristics curve was used for estimating the under the curve.

DETAILED DESCRIPTION:
Diagnosis of periodontal diseases and conditions was arranged according to the radiographic and clinical diagnostic criteria proposed by the 2017 World Workshop on Classifcation of Periodontal and Peri-implant Diseases and Conditions; 20 patients with Stage III Grade B generalized periodontitis , 20 patients with Stage III Grade C generalized periodontitis , 19 gingivitis patients and periodontally healthy volunteers were included in this study.

The clinical periodontal examination of the healthy and periodontitis subjects consisted of plaque index (PI), probing pocket depth (PPD), clinical attachment level (CAL), and bleeding on probing (BOP) recorded. CAL was calculated by adding GR to the PPD values. Averages for full mouth PPD, CAL, and the percentage of sites with BOP were calculated for each subject. A single calibrated examiner (VO) conducted a full mouth periodontal examination of all participants. The measurements were performed using a Williams periodontal probe (Hu-Friedy, Chicago, IL, USA). All measurements were performed full mouth and at 4 sites (mesio-buccal, mid-buccal, distobuccal, and mid-lingual) for each tooth. Before clinical measurements, intra-examiner calibration was performed by measuring PPD and CAL values twice on five patients with one day interval resulting in intraclass correlation coefficients were 0.92 for PD and 0.90 for CAL.

GCF samples were taken from the buccal aspects of two nonadjacent interproximal sites in single-rooted teeth. In periodontitis groups, GCF was sampled from two deepest pockets of single-rooted teeth. Samples were collected from the sites with visible signs of inflammation in gingivitis group and without BOP in the healthy group. The selected areas were carefully cleared of supragingival plaque using sterile curettes, isolated with cotton rolls, and slightly air-dried to avoid contamination.

Standardized filter paper strips (PerioPaper, Proflow, Amityville, NY) were used for GCF sampling. Sterile paper strips were gently inserted into the gingival sulcus or pocket until mild resistance was felt and left there for 30 seconds. Mechanical irritation was avoided and strips visually contaminated with blood were discarded. A precalibrated electronic device measured the absorbed fluid volume (Periotron 8010, Oraflow, Amityville, NY). The readings were converted to an actual volume (microliter, μL) by reference to the standard curve. The paper strips were individually placed into a sterile polypropylene tube and stored at -80◦C for further analysis.

Annexin-A1 levels were studied with commercially available kits using the ELISA method (Bioscience SRB, catalog no: 201-12-3158). The optical density was measured spectrophotometrically at a wavelength of 450 nm (Tecan). The assay ranges for the Annexin-A1 kit were 0.20-20 ng/mL, sensitivity 0.2 ng/mL, and the intra- and interassay coefficients of variance (CV%) were<10%. The results were presented as ng.

Carbonic anhydrase 1 levels were studied with commercially available kits using the ELISA method (Bioscience SRB, catalog no: SRB-T-88927). The optical density was measured spectrophotometrically at a wavelength of 450 nm (Tecan). The assay ranges for the CA I kit were 3.12-200ng/mL, sensitivity <1.875ng/mL, and the intra- and interassay coefficients of variance (CV%) were<10%. The results were presented as ng.

EEF1G levels were studied with commercially available kits using the ELISA method (Bioscience SRB, catalog no: 201-12-3732). The optical density was measured spectrophotometrically at a wavelength of 450 nm (Tecan). The assay ranges for the EF1- Ɣ kit were 31.25-2000pg/mL, sensitivity <12.4pg/mL, and the intra- and interassay coefficients of variance (CV%) were<10%. The results were presented as ng.

Statistical analysis was performed using non-parametrical techniques. Comparisons between the study groups were performed using the Kruskal-Wallis test. When there were significant differences (p < 0.05), post-hoc 2-group comparisons were assessed with Bonferroni-corrected Mann-Whitney U tests, and p-values < 0.05 was considered significant. All data analysis was performed using a statistical package (Abacus Concepts Inc., Berkeley, CA, USA). The diagnostic accuracy, sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), receiver operating characteristic (ROC) curve, and area under the ROC curve (AUC) of the test dataset were assessed. P values < 0.05 were considered statistically significant, and 95% confidence intervals (CIs) were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers with no history of smoking(determined by self-reporting)
* Individuals who had at least 20 teeth(exclude wisdom teeth)

Exclusion Criteria:

* Pregnant and lacting women
* Patients who under any medication including immunosuppressants, steroids, non-steroidal anti-inflammatory drugs, antibiotics, antiepileptic drugs, calcium channel blockers, beta,blockers, anticoagulants, hormonal contraceptives and nutritional supplements within 6 monthsi topical antiseptic solutions in the last 3 months.
* Patients with diagnosed medical illness such as diabetes mellitus, rheumatoid arthritis, cardiovascular diseases, immunological diseases.

Ages: 20 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 80 systemically healthy and non-smoker individuals(39 males, 41 females) aged 20-61 years were consecutively included.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2022-12-16 (Actual)

PRIMARY OUTCOMES:
Gingival crevicular fluid Annexin-A1 levels | 24 hours after clinical periodontal measurements
  ng
Gingival crevicular fluid Carbonic Anhydrase-1 levels | 24 hours after clinical periodontal measurements
  ng
Gingival crevicular fluid Elongation Factor-1 Gamma- Ɣ levels | 24 hours after clinical periodontal measurements
  ng

CONTACTS AND LOCATIONS:
Overall Officials: Bilge Cansu Uzun Saylan, Principal Investigator — Dokuz Eylul University; Veli Özgen Öztürk, Principal Investigator — Aydin Adnan Menderes University; Harika Atmaca İlhan, Principal Investigator — Manisa Celal Bayar University; Gülnur Emingil, Study Director — Ege University
Locations (1):
- Dokuz Eylul University, Faculty of Dentistry, Department of Periodontology, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided